CLINICAL TRIAL: NCT03519646
Title: Evaluation of the Safety in the Combination Usage of Cerdelga and Cerezyme in Type III Gaucher Disease Patients and the Efficacy on Soft Tissue Diseases.
Brief Title: Eliglustat on Gaucher Disease Type IIIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201612250MIPB
Record Dates: First submitted 2018-03-20; First posted 2018-05-09 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2021-01

CONDITIONS: Gaucher Disease, Type III
Keywords: Enzyme Replacement Therapy; Eliglustat (Cerdelga®)
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental Case_Eiglustat (Experimental): Besides regular ERT, patients also need to take Eiglustat for 24 months.
  Interventions: Drug: Eliglustat

INTERVENTIONS:
Drug: Eliglustat — 1. This is a 3-year study and the enrollment time of this study is 24 months.
  2. The participants have to receive the investigational agent, Cerdelga
  3. The participants have to go back to the hospital and receive the investigational agent and take the test before receving Cerdelga, and 2 weeks, 1, 3, 6, 12, 18 and 24 months after receiving Cerdelga.
  4. IMP Administration Method: Cerdelga have 21 mg、42 mg and 84 mg capsule.
  5. No need for fasting before use, but can't take with grapefruit juice.
  6. Five ml Blood and 10 ml urine shoud be taken before receiving Cerdelga, and 1, 3, 6, 12, 18 and 24 months after receiving Cerdelga for Gaucher related biomarkers test.
  Other Names: Cerdelga

SUMMARY:
Evaluation of the safety in the combination usage of Cerdelga and Cerezyme in type III Gaucher disease patients and the efficacy on soft tissue diseases.

DETAILED DESCRIPTION:
* This is a 3-year study and the enrollment time of this study is 24 months.
* The participants have to receive the investigational agent:Cerdelga.(Cerdelga have 21 mg、42 mg and 84 mg capsule.)
* The participants have to go back to the hospital and receive the investigational agent and take the Gaucher related biomarkers test before receiving Cerdelga, and 2 weeks, 1, 3, 6, 12, 18 and 24 months after receiving Cerdelga.
* The participants have to inform if any adverse events happened.
* The investigators will follow up by phone if adverse events happened in the participants after one months start the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Gaucher disease patients diagnosed by low B-glucocerebrosidase deficiency and GBA mutation .
* The participant is at least 6 years old at time of enrollment.
* Under stable Cerezyme dosage for at least for 3 months.
* Presence of lymphadenopathy.
* Patient (and/or their parent/legal guardian) is willing to participate and able to provide signed informed consent.

Exclusion Criteria:

* The participant is CYP2D6 ultra-rapid metabolizer.
* The participant had received substrate reduction therapy for Gaucher disease within 3 months of enrollment.
* The participant had any clinically significant disease other than GD, including cardiovascular (especially arrhythmia), renal, liver, pulmonary, endocrinopathy, hypokalemia, or hypomagnesemia that may confound the study result.
* The participant is pregnant or lactating.
* The participant is known to be allergy to Cerdelga.
* The participant use drugs that will strongly inhibit CYP2D6 or CYP3A activity .

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From date of enrollment with information consent form until 24 months or date of death from any cause, whichever came first.
  Number of adverse events in patients.

SECONDARY OUTCOMES:
Assessment of Gaucher related biomarkers test :CCL18 (30% decrease) | Baseline,1,3,6,12,18 and 24 months after receiving Cerdelga.
  Measure of Gaucher disease type I biomarkers:CCL18(ng/ml) in plasma.
Assessment of Gaucher related biomarkers test :Lyso GL1(30% decrease) | Baseline,1,3,6,12,18 and 24 months after receiving Cerdelga.
  Measure of Gaucher disease type I biomarkers:Lyso GL1 (ng/mL) in plasma
Assessment of Gaucher related biomarkers test:Chitotriosidase(30% decrease) | Baseline,1,3,6,12,18 and 24 months after receiving Cerdelga.
  Measure of Gaucher disease type I biomarkers:Chitotriosidase(nmol/ml/h) in plasma.
Change in lymphadenopathy manifestations. | From date of enrollment with information consent form until 24 months or date of death from any cause, whichever came first.
  Physician will pay close attention to the lymphadenopathy including size, location, and number of enlarged lymph nodes, evaluate by palpation and radiological (MRI examination). The total size of the lympadenopathy will be combined into one report as "Total size" cm^3.
Pharmacokinetics | Plasma concentration-time data will be obtained pre-dose (within 30 minutes prior to dosing) and at 1, 2, 6, 12, 26, 36 hours after 1st dosing, and 1,3,6,12,18 and 24 months thereafter.
  Eliglustat plasma concentration over time

CONTACTS AND LOCATIONS:
Overall Officials: Ni-Chung Lee, M.D., Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan